CLINICAL TRIAL: NCT04980768
Title: Association of Apical Periodontitis With Systemic Levels of Hs-CRP and Hemogram Indices: A Clinical Study.
Brief Title: Association of Apical Periodontitis With Hs-CRP and Hemogram Indices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP & Systemic Markers
Record Dates: First submitted 2021-07-04; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Periapical Periodontitis
Keywords: Apical periodontitis; hsCRP; root canal treatment; hemogram; inflammation
MeSH Terms: conditions — Periapical Periodontitis; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Root canal treatment (Other): Root canal treatment will be provided to all the participants with the diagnosis of apical periodontitis.
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Root canal treatment — Patients with apical periodontitis will undergo root canal treatment.

SUMMARY:
There is lack of evidence on resolution of signs of systemic inflammatory markers by successful elimination of periapical inflammation by endodontic treatment. Complete blood count (CBC) may have potential to detect various inflammatory conditions but its use for this purpose is sparsely reported. To the best of our knowledge effect of chronic apical periodontitis on various parameters of complete blood count has not been studied.

DETAILED DESCRIPTION:
Prevalence of Apical periodontitis (AP) is reported in the range of 17% to 65% with higher prevalence reported in older patients. Infection of the pulp tissue of the affected tooth is the principal cause of apical periodontitis and it is characterised by inflammation of the periradicular tissues. Presentation of AP varies from classical signs of inflammation (pain, swelling, loss of function) to being completely asymptomatic with only signs of apical bone resorption on the radiograph. Histological changes seen in AP is localized infiltration of inflammatory cells and bone resorptions. AP can be treated by root canal treatment (RCT) which comprises elimination of microbes and their toxic products followed by filling of the root canal by an inert material. It also acts to limit the spread of microbial infection seen in AP to jaw and the other parts of the body.

Apical periodontics if left untreated can cause serious complications. Infection and loss of function caused by loss of teeth may jeopardize overall health of the patients. Chronic infection like untreated AP may also influence development and progression of other serious conditions. Numerous inflammatory mediators are responsible for eliciting inflammatory reactions seen in AP for example both IL-1beta and TNF-alpha are found in periapical lesions and IL-1beta is suggested to cause greater bone resorption in patients of AP. Role of these mediators in AP is to cause vasodilation, increased vascular permeability and recruit other inflammatory cells. It is also been suggested that increased inflammatory mediators seen in AP may also enhance the systemic inflammation. Inflammation induced tissue damage may vary in different disease, however the markers that trigger this damage are very similar. They all act to increase the rate of the inflammatory process, cause tissue destruction and may even be involved in development of clinical symptoms. For example, markers like hsCRP is associated with various steps of atherogenesis and is also found elevated in AP. Studies have reported significantly higher levels of endothelial dysfunction in patients of apical periodontitis which were found to reduce to normal level following root canal treatment.

A recent systematic review has found significant difference in levels of CRP and IL-6 in AP subjects than control. IL-6 plays role in initiation of autoimmune disease and chronic inflammation and also contributes in low grade systemic inflammation. The same systematic review and meta-analysis has found only eight interventional study that studied effect on inflammatory marker before and after treatment. The data from these studies were also heterogenous with wide variety of treatment reported. Only two studies are available which has evaluated effect of endodontic treatment on levels of isolated groups of inflammatory mediators and stress markers like reactive oxygen species and circulatory immune complex. TNF- α is indicated to be responsible for adverse pregnancy outcome and along with CRP may enhance the insulin resistance. Similarly, complete hemogram indices like mean platelet volume, neutrophil-lymphocyte ratio is altered in chronic inflammatory conditions and their estimation could be useful in evaluating overall systemic inflammatory burden of patients of AP. To the best of our knowledge no study so far has evaluated effect of non-surgical root canal treatment on the levels of hsCRP and complete hemogram parameters. Therefore, this study proposes to compare these markers in patients of AP and healthy control and also before and two years after root canal treatment.

Medical and Dental Examination Prior to treatment a detailed medical and dental history will be recorded. Oral clinical examinations will include hard and soft tissue evaluation. Pulp sensibility test will be carried out along with percussion and palpation of the affected tooth. The periapical radiographic examinations will be carried out at standard exposure parameters to detect apical bone resorption. Periodontal clinical parameters will be evaluated at 6 sites in all teeth, including probing depths (PDs), the clinical attachment level, and bleeding on probing at the base of the crevice, excluding third molars. The periodontal assessment will be made with a manual periodontal probe (UNC 15; Hu-Friedy, Chicago, IL).

Blood Samples and Laboratory Analysis Fasting blood samples will be obtained by venipuncture of the ante-cubital vein. Blood sample will be submitted to the clinical laboratory of the Department of Biochemistry PGIMS and Department of Oral Pathology, PGIDS, Rohtak, Haryana for the quantitative analysis of hs-CRP and complete hemogram analysis respectively.

Technique for ELISA: Whole blood sample will be kept at 4°C overnight and centrifuged for 15 minutes at approximately 6000 rpm. Serum will be separated and stored in aliquots at -80 °C in the until use. Serum hsCRP assay kit will be used. ELISA is a sandwich enzyme immunoassay. A monoclonal antibody specific for these markers will be pre- coated on the microplate. Standard and sample will be pipetted into wells and any marker present will be bound by immobilized antibody. After washing away any unbound substances, enzyme- linked polyclonal antibody specific for hs-CRP will be added to the wells.

After an incubation period amplifier solution will be added to the wells, and the color will develop in proportion to the amount of hsCRP bound in the initial stage. The intensity of the color will be measured.

Root Canal treatment Access opening will be done after rubber dam isolation and administration of local anesthesia. debridement of the pulp chamber will be done and all canal orifices will be identified. Negotiation of canals will be done. Working length will be determined using root ZX apex locator and will be verified radiographically. Coronal enlargement will be done using Gates- Glidden drills. The apical third of the root canal will be instrumented up to size 35 for mesial and up to size 45 for distal canals. Finally, root canals will be further instrumented with step-back technique enlargement in 1 mm increments to 3 sizes larger than the master apical file. Irrigation will be carried out using 5 mL of a 5% NaOCl solution between files. After preparation, the root canals will be irrigated with 5 mL 17% EDTA for 3 minutes to remove smear layer, followed by 5 mL 5% NaOCl. The final irrigation will be done with 5 mL distilled water. The root canals will be dried using paper points and filled with laterally condensed gutta-percha (Dentsply Maillefer) and Zinc oxide Eugenol based sealer mixed according to manufacturers' instructions. Gutta- percha will be cut with a heated instrument and vertically condensed right at the orifice opening of the canals. Final composite resin restoration will be done following manufacturer instruction.

Follow up Follow up and clinical and radiographic examination will be carried out at six months. Re-assessment of hs-CRP and complete hemogram indices will also be done of all patients at 6 months

ELIGIBILITY:
Inclusion Criteria:

* Pulpal necrosis in mature mandibular molar as confirmed by negative response to pulp sensibility test (cold and electric pulp test)
* Radiographic evidence of apical periodontitis in the form of periapical radiolucency
* Radiographic alveolar bone breakdown not more than one third of root length.

Exclusion Criteria:

* Obese (BMI >30 kg/m2), smoker, pregnant, diabetic, immunocompromised or have any other systemic inflammatory condition.
* Having a positive history of antibiotic use within the past month or require antibiotic premedication for dental treatment (including infective endocarditis or prosthetic joint prophylaxis).
* Teeth having previous root fillings, unrestorable teeth, fractured/perforated roots, grade 3 mobility, and history of recent periodontal therapy (within previous 6 months).
* Teeth with established endodontic-periodontal lesions exhibiting <2 mm radiopaque bone between the root apex.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Level of hs-CRP | Baseline-3 months
  Serum level of hs-CRP will be measured using ELISA in g/dl.
Hemogram indices | Baseline-3 months
  Complete hemogram parameters in percentage will be assessed using automated machine.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Haryana, India